CLINICAL TRIAL: NCT04850599
Title: A Single-Arm Phase II Study of Isatuximab With Carfilzomib and Pomalidomide in Relapsed or Refractory Multiple Myeloma
Brief Title: Isatuximab, Carfilzomib, and Pomalidomide for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Rebecca W. Silbermann, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021808; NCI-2021-02297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021808 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; isatuximab; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (isatuximab, carfilzomib, pomalidomide) (Experimental): Patients receive isatuximab IV over 30-60 minutes on days 1, 8, 15, and 22 of cycle 1, and days 1 and 15 of subsequent cycles, carfilzomib IV over 10 to 30 minutes on days 1, 8, 15, and pomalidomide PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Biological: Isatuximab; Drug: Pomalidomide

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Biological: Isatuximab — Given IV
  Other Names: Hu 38SB19; Isatuximab-irfc; SAR 650984; SAR650984; Sarclisa
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies the effect of isatuximab, carfilzomib, and pomalidomide in treating patients with multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Isatuximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as pomalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving isatuximab, carfilzomib, and pomalidomide may help treat patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the rate of response following treatment with isatuximab combined with carfilzomib and pomalidomide (isatuximab [Isa] carfilzomib [Car] pomalidomide [Pom]).

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of the IsaCarPom combination. II. To assess duration of disease response following treatment with the IsaCarPom regimen.

III. To assess depth of IsaCarPom treatment as it relates to timing of subsequent therapies.

IV. To assess progression-free survival associated with IsaCarPom. V. To assess overall survival associated with IsaCarPom.

EXPLORATORY OBJECTIVE:

I. To molecularly assess the depth of IsaCarPom treatment by measuring minimal residual disease (MRD).

OUTLINE:

Patients receive isatuximab intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 22 of cycle 1, and days 1 and 15 of subsequent cycles, carfilzomib IV over 10 to 30 minutes on days 1, 8, 15, and pomalidomide orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative (LAR) must provide written informed consent before any study specific procedures or interventions are performed
* Participants must be >= 18 years of age
* Histologically or cytologically confirmed diagnosis of multiple myeloma (MM) as defined by 2016 International Myeloma Working Group (IMWG) criteria
* Relapsed or relapsed and refractory (R/R) MM, as defined by International Myeloma Working Group (IMWG) criteria:

  * Relapsed myeloma: Previously treated myeloma that has progressed and is neither "refractory myeloma" nor "relapsed-and-refractory myeloma"
  * Refractory myeloma: Nonresponsive myeloma while on primary or salvage therapy, or progresses within 60 days of last therapy. Nonresponsive disease is defined as failure to achieve minimal response (MR) or better, achieved with any therapy. Cases in which there is no significant change in M protein and no evidence of clinical progression, are included, as well those cases that progress in disease course

    * Primary refractory myeloma: Disease that is nonresponsive in patients who have never achieved a minimal response or better with any therapy
    * Relapsed-and-refractory myeloma: Disease that is nonresponsive while on salvage therapy or progresses with 60 days of last therapy after achieving MR or better previously before progressing
* Participant has received at least 1 line of prior therapy.

  * Prior exposure to proteasome inhibitor is permitted. The washout period is 2 weeks (14 days) prior to start of study treatment (cycle 1 day 1 [C1D1])
  * Prior exposure to immunomodulatory imide drug (IMiD) therapy (lenalidomide, pomalidomide, or thalidomide) is permitted. The washout period is 2 weeks (14 days) prior to start of study treatment (C1D1)
  * Prior treatment with anti-CD38 therapy (e.g., daratumumab) is permitted. The washout period is 6 months prior to start of study treatment (C1D1)
* Measurable disease with at least one of the following:

  * Monoclonal immunoglobulin spike on serum protein electrophoresis of >= 0.5 g/dL
  * Urine monoclonal immunoglobulin spike of >= 200 mg/24 hours
  * Involved free light chain (FLC) >= 10 mg/dL and an abnormal serum FLC ratio (i.e., < 0.26 or > 1.65)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Toxicity related to prior therapies that, in the opinion of the investigator, would potentially be worsened with anti-CD38 therapy should be resolved to baseline or less than grade 1
* Anticipated life expectancy of at least 6 months (per investigator discretion)
* No contraindication to receiving thromboprophylaxis for pomalidomide
* Patients must have normal marrow and organ function as defined by:

  * Absolute neutrophil count (ANC) ≥ 1,000/uL. Patients may receive growth factor support to meet screening criteria. Screening ANC must be redrawn 72 hours after growth factor dosing. Screening platelets or hemoglobin must be redrawn 72 hours after transfusion
  * Platelets >= 75,000/uL within 14 days prior to registration. Patients may have received transfusion if > 7 days prior to registration
  * Hemoglobin concentration of >= 8.0 g/dL within 14 days prior to registration. Patients may have received transfusion if greater than 7 days prior to registration
  * Must have adequate liver function, as defined by:

    * Normal total bilirubin (as per institutional upper limits of normal [IULN]), except if due to Gilbert's syndrome, or other documented historical elevations in serum bilirubin levels, at the discretion of the investigator, AND
    * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2 x IULN
  * Must have adequate renal function, as defined by:

    * Creatinine clearance (CrCl) of >= 30 mL/min, as measured by a 24-hour urine collection or as estimated by the Cockcroft and Gault formula. The serum creatinine value used in the calculation must have been obtained within 35 days prior to registration.
    * For patients with a creatinine clearance within the range of 30-45 mL/min, stability (i.e., not deteriorating) must be demonstrated over a period of 8 weeks prior to enrollment in the study
  * Lab parameters must continue to be met at the time of registration. If parameters not met at the intended C1D1, transfusion or growth factor support may be considered in consultation with the team, if the individual is still within the screening window
* Left ventricular ejection fraction (LVEF) by echocardiogram >= 40%. The echocardiogram study should be obtained during screening or up to 60 days prior to consent
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to receiving the first dose of study medication. If the urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female participants of childbearing potential (FOCBP) must agree to use highly-effective method(s) of contraception during the study and for 3 months after the last dose of study drug. FOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study drug

Exclusion Criteria:

* Waldenstrom macroglobulinemia
* Multiple myeloma of immunoglobulin M (IgM) subtype
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia (> 2.0 x 10^9/L circulating plasma cells by standard differential)
* Myelodysplastic syndrome
* Participants with known or suspected amyloidosis
* Individuals that are refractory to prior treatment with either carfilzomib or pomalidomide
* Intolerance leading to discontinuation of either carfilzomib or pomalidomide
* Prior allogeneic stem cell transplant
* Second malignancy requiring concurrent treatment or those with non-hematological malignancies (except non-melanoma skin cancers). Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the principal investigator (PI). Cancer treated with curative intent > 5 years previously is allowed
* Any known allergies or hypersensitivity to isatuximab or other monoclonal antibody therapies and required premedications
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Hypersensitivity to any of the components of study therapy that is not amenable to premedication with steroids and H2 blockers
* Participant has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, of the first dose of study medication. Wash-out period of prior anti-CD38 therapy (e.g. Daratumumab) is 6 months before first dose of study medication.

  * Exception: Emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 mg per day for a maximum of 4 days) before treatment is not a barrier to eligibility
* Participant has undergone autologous stem cell transplant within 90 days of the first dose of study medication
* Ongoing adverse events related to a previously administered anti-myeloma therapy (including radiation therapy) >= grade 1

  * Exception: Potential participants with =< grade 2 neuropathy may, at the discretion of the investigator, qualify for the study
* Active autoimmune disease, except vitiligo or hypothyroidism
* Active and ongoing steroid use, except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, chronic obstructive pulmonary disease [COPD], allergic rhinitis, or dermatologic conditions) and the emergency use of corticosteroids outlined above
* Known human immunodeficiency virus (HIV) infection
* Ongoing or active systemic infection
* Seropositive for hepatitis B virus (HBV) defined by a positive test for hepatitis B surface antigen (HBsAg). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. Exception: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Seropositive for hepatitis C virus (HCV) (except in the setting of a sustained virologic response, defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV), pulmonary hypertension, unstable angina, or myocardial infarction within the past 6 months
* Participant has received a live vaccine within 30 days of planned start of study therapy
* A history of non-infectious pneumonitis that required treatment with steroids, or current pneumonitis
* Diagnosis of immunodeficiency or treatment with any form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Pregnant or breastfeeding
* Any medical or psychiatric conditions that in the opinion of the PI would preclude safe participation in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2029-02-21 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to end of cycle 4 (each cycles is 28 days), disease progression, start of new anti-myeloma therapy, or death (whichever occurs first)
  Defined as the proportion of participants who achieve a response >= partial response (PR) (i.e., PR, very good partial response, complete response, or stringent complete response) according to International Myeloma Working Group criteria. ORR will be measured from start of study treatment (i.e., cycle 1 day 1) to the earliest of the following events: end of cycle 4, start of new anti-myeloma therapy, documented disease progression, or death. Will be evaluated using the response-evaluable analysis set. A point estimate and exact 95% confidence interval will be provided.

SECONDARY OUTCOMES:
Incidence of grade > 2 toxicities | Up to 30 days after discontinuing study treatment
  Evaluated per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Descriptive statistics will be used to summarize all on-study adverse events (AEs), grade 3-4 AEs, treatment-related AEs, grade 3-4 treatment-related AEs, SAEs, treatment-related severe (S)AEs, and AEs leading to study therapy discontinuation. Grade 3-4 laboratory abnormalities will be summarized using worst grade NCI CTCAE v5.0 criteria.
Duration of response (DOR) | From initial disease response (>= PR) until disease progression, disease-related death, death from other cause (competing risk), or end of follow-up (censored), whichever occurs first, assessed up to 24 months
  Defined for participants with a confirmed response (>= PR) as the time between first documentation of response and disease progression according to IMWG criteria or death due to disease, whichever occurs first. Will be analyzed using the response-evaluable analysis set. Since non-progression, non-multiple myeloma (MM)-related death is a competing risk when assessing DOR, this endpoint will be estimated by cumulative incidence functions (one for progression or MM-related death, one for non-progression death) and modeled with Fine-Gray sub-distribution hazard regression.
Time to next treatment | From start of study regimen until start of new anti-myeloma therapy, death from any cause before new therapy, or end of follow-up (censored), whichever occurs first, assessed up to 24 months
  Will be estimated by the Kaplan-Meier method and modeled with Cox regression.
Progression-free survival | From start of study treatment until disease progression, death, or end of follow-up (censored), whichever occurs first, assessed up to 24 months
  Will be analyzed using the response-evaluable analysis set. Will be estimated by the Kaplan-Meier method and modeled with Cox regression.
Overall survival | From start of study treatment until death or last known alive (censored), assessed up to 24 months
  Will be estimated by the Kaplan-Meier method and modeled with Cox regression.

OTHER OUTCOMES:
Frequency of minimal residual disease negative remissions at time of complete response | First post-baseline bone marrow or aspirate until last standard of care bone marrow biopsy on study (including follow-up), assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca W Silbermann, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States